CLINICAL TRIAL: NCT03578692
Title: Clinical Value of Inflammation-related Indicators of Blood and Fecal Calprotectin in Predicting the Surgery Rate of Acute Severe Ulcerative Colitis
Brief Title: Indicators Predicting Surgery in Acute Severe Ulcerative Colitis(ASUC)
Status: Completed | Type: Observational
Sponsor: Gao Tao (Other)
Responsible Party: Sponsor-Investigator, Gao Tao, Clinical Professor, Nanjing PLA General Hospital
Organization: Nanjing PLA General Hospital (Other)
Other Study IDs: 2018NLY052
Record Dates: First submitted 2018-05-07; First posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Ulcerative Colitis Acute; Surgery
Keywords: acute severe ulcerative colitis; predictive indicator; surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery group: The protocol for patients assigned to surgery group was as follows. ASUC patients were admitted in, estimated their baseline situations and tested their blood and fecal indicators including PCT, IL-6 and FC on admission. All patients were treated according to the ECCO guideline 2012. Patients who showed bad response to medicine (glucocorticoid for 5 days and rescue therapy for 3 days) were recommended and classified in the surgery group. Their baseline manifestations were collected and compared with the medical group, to exploit the baseline indicators with great sensitive and specificity predicting the high risk for surgery.
- Medical group: The protocol for patients assigned to medical group was as follows. ASUC patients were admitted in, estimated their baseline situations and tested their blood and fecal indicators including PCT, IL-6 and FC on admission. All patients were treated according to the ECCO guideline 2012. Patients who showed response to medicine (glucocorticoid for 5 days or rescue therapy for 3 days) were classified in the medical group. Their baseline manifestations were collected and compared with the surgery group.

SUMMARY:
Acute severe ulcerative colitis [ASUC] patients have high risk of no response to medical treatments and might miss the best timing for surgery when waiting for the medical response. Thus, we investigated whether biomarkers which could early predict the surgery risk of patients with ASUC on admission.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criterion was patients clearly diagnosed as acute severe ulcerative colitis.

Exclusion Criteria:

Patients younger than 18 years-of-age, complicated with malignancy in colon and pregnant were excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All acute severe ulcerative colitis patients were admitted in hospital and prospectively followed during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Colon operation | 30 days
  100% direct approximation of inevitable surgery

SECONDARY OUTCOMES:
No response to medical treatments | 5 days
  Medical treatments involve glucocorticoids, Immunosuppressant and biologicals for ulcerative colitis. The Oxford Index measured everyday, consisting of CRP and stool frequency, is used to evaluate the response to the treatment. If the Oxford Index does not reduce after 5-day medical treatment, this situation is deemed as no response to medical treatment
30-day mortality | 30 days
  All-cause mortality within 30 days